CLINICAL TRIAL: NCT05689840
Title: Association Between Post-covid Infection Status and Perioperative Morbidity: A Ambispective Cohort Study
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K23C0257
Record Dates: First submitted 2023-01-18; First posted 2023-01-19 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Complication of Anesthesia; Complication of Surgical Procedure; Complication,Postoperative; Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 0-1 week group: Patients who have been infected with Covid-19 with 0-1 week post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- 1-2 weeks group: Patients who have been infected with Covid-19 with 1-2 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- 2-3 weeks group: Patients who have been infected with Covid-19 with 2-3 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- 3-4 weeks group: Patients who have been infected with Covid-19 with 3-4 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- 4-5 weeks group: Patients who have been infected with Covid-19 with 4-5 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- 5-6 weeks group: Patients who have been infected with Covid-19 with 5-6 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention
- over 6 weeks group: Patients who have been infected with Covid-19 with over 6 weeks post-COVID interval before surgery.
  Interventions: Procedure: Receiving inpatient surgical intervention

INTERVENTIONS:
Procedure: Receiving inpatient surgical intervention — Receiving inpatient surgical intervention in Peking Union Medical College Hospital

SUMMARY:
With the knowledge of currently transmitted omicron variant being less virulent, over 90 percent of the Chinese population is fully vaccinated, and the Chinese health workers have sufficient experience treating the illness. China 's epidemic prevention and control has entered a new stage to restore the normal functioning of society and basic medical services, On Dec, 7, China released a circular on further optimizing its COVID-19 response, announcing 10 new prevention and control measures.This has marked the watershed for sharply increased number of elective surgical patients diagnosed with COVID-19 during preoperativley, fully recovered or during recovery.

Beijing faced a wave of omicron infection starting that would result in of a wide range of population infections. At which time there is limited evidence regarding the optimal timing of surgery following SARS-CoV-2 infection especially for omiron among Chinsese patients .This study intends to explore the relationship between the incidence of postoperative complications after elective surgery and COVID-19 infection in Peking Union Medical College Hospital, and provide data support for the policy formulation of elective surgical timing for patients after COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. All patients having pre-operative SARS-CoV-2 infection diagnosis Dec 1st 2022 to Feb 28th 2023.

[The COVID-19 diagnosis is based on either (a) a positive RT-PCR nasopharyngeal swab, (b) positive antigen rest before surgery, or (c) clinical diagnosis made before surgery].

Exclusion Criteria:

1. Patients diagnosed with SARS-CoV-2 infection on the day of surgery or during postoperative days.
2. Day surgery or outpatient surgery.
3. Patients unwilling to participate or provide COVID-19-related information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the part of retrospective study，the investigators intend to include patients who had pre-operative SARS-CoV-2 infection diagnosis and received inpatient surgical intervention at Peking Union Medical College Hospital from December 1, 2022 to January 8, 2023.
  For the part of prospective study，the investigators intend to include patients who will receive inpatient surgical intervention with pre-operative SARS-CoV-2 infection diagnosis at Peking Union Medical College Hospital from January 9, 2023 to February 28, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | During the procedure
  The composite primary outcome included pulmonary complications (pneumonia, acute respiratory distress syndrome, or acute respiratory failure, reintubation, unplanned use or prolongation of postoperative mechanical ventilation), cardiovascular complications (deep vein thrombosis, pulmonary embolism, myocardial infarction, newly onset arrhythmia, ischemic stroke, and acute kidney injury), and infectious complications other than pulmonary infection (urinary tract infection, surgical site infection, and sepsis).

OTHER OUTCOMES:
Length of hospital stay | Immediately after discharge
  Calculate the number of days the patient stays in the hospital.
Readmission rate during 30 days after surgery | 30 days after operation
  Readmission due to surgery complications during 30 days after operation
Postoperative mechanical ventilation time | During the procedure
  Length of mechanical ventilation time after surgery
Mortality after operation | 1 month, 3 months, 6 months, 12 months after operation
  Mortality after operation in 1 month, 3 months, 6 months, 12 months
Intraoperative respiratory complication | During the surgery
  Intraoperative respiratory complication: a composite of intraoperative bronchospasm, poor oxygenation, and reintubation.
the WHODisability Assessment Schedule (WHODAS 2.0) | 6 months after operation
  * Step 1-Summing of recoded item scores within each domain.
  * Step 2-Summing of all six domain scores.
  * Step 3-Converting the summary score into a metric ranging from 0 to 100 (where 0=no disability; 100=full disability).
Brief Pain Inventory (BPI) | 6 months after operation
  Brief Pain Inventory used to assess the intensity of pain

CONTACTS AND LOCATIONS:
Overall Officials: Shen Le, PhD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Boghdadly K, Cook TM, Goodacre T, Kua J, Denmark S, McNally S, Mercer N, Moonesinghe SR, Summerton DJ. Timing of elective surgery and risk assessment after SARS-CoV-2 infection: an update: A multidisciplinary consensus statement on behalf of the Association of Anaesthetists, Centre for Perioperative Care, Federation of Surgical Specialty Associations, Royal College of Anaesthetists, Royal College of Surgeons of England. Anaesthesia. 2022 May;77(5):580-587. doi: 10.1111/anae.15699. Epub 2022 Feb 22. PMID 35194788
- [Background] COVIDSurg Collaborative. Outcomes and Their State-level Variation in Patients Undergoing Surgery With Perioperative SARS-CoV-2 Infection in the USA: A Prospective Multicenter Study. Ann Surg. 2022 Feb 1;275(2):247-251. doi: 10.1097/SLA.0000000000005310. PMID 34793350
- [Background] Quinn KL, Huang A, Bell CM, Detsky AS, Lapointe-Shaw L, Rosella LC, Urbach DR, Razak F, Verma AA. Complications Following Elective Major Noncardiac Surgery Among Patients With Prior SARS-CoV-2 Infection. JAMA Netw Open. 2022 Dec 1;5(12):e2247341. doi: 10.1001/jamanetworkopen.2022.47341. PMID 36525270
- [Background] Bryant JM, Boncyk CS, Rengel KF, Doan V, Snarskis C, McEvoy MD, McCarthy KY, Li G, Sandberg WS, Freundlich RE. Association of Time to Surgery After COVID-19 Infection With Risk of Postoperative Cardiovascular Morbidity. JAMA Netw Open. 2022 Dec 1;5(12):e2246922. doi: 10.1001/jamanetworkopen.2022.46922. PMID 36515945
- [Derived] Che L, Yu J, Jin D, Bai X, Wang Y, Zhang Y, Xu L, Shen L, Huang Y. Impact of previous COVID-19 infection on postoperative complications and functional recovery: a 1-year follow-up ambispective cohort study. Int J Surg. 2025 Jan 1;111(1):481-491. doi: 10.1097/JS9.0000000000001869. PMID 38935110
- [Derived] Che L, Yu J, Bai X, Wang Y, Zhang Y, Xu L, Shen L, Huang Y. Association between post-COVID-19 status and perioperative morbidity and mortality: protocol for an ambispective cohort study. BMJ Open. 2023 Sep 14;13(9):e074337. doi: 10.1136/bmjopen-2023-074337. PMID 37709339